CLINICAL TRIAL: NCT05882695
Title: A Phase 1/2a, Randomized, Double Blind, Placebo Controlled, Single and Multiple Dose Escalation Study in Healthy Volunteers and an Expansion Cohort in Adult Participants With Amyotrophic Lateral Sclerosis (ALS) to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SPG302
Brief Title: Study of SPG302 in Healthy Volunteers and ALS Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spinogenix (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPG302-ALS-001
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; regenerative; synapse
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Phase 1 randomized, double-blind, placebo-controlled, single, and multiple ascending dose study in HV and a repeat dose expansion in ALS cohort(s)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Experimental Part 1: Active SPG302 to be administered to healthy volunteers (SAD) (Experimental): 8 participants will be randomized in a 3:1 ratio to active or placebo. Study intervention will be administered orally once. Randomization to each SAD cohort will be done in a staggered manner; initially 2 sentinel participants (1 active and 1 placebo) will be randomized and dosed and after a safety evaluation period after the dose without clinically significant adverse events (AEs) and investigator approval, then, 6 additional participants will be randomized and dosed (5 active and 1 placebo) at the discretion of the Investigator according to the randomization schedule
  Interventions: Drug: SPG302
- Placebo Comparator Part 1: Placebo comparator to be administered to healthy volunteers (SAD) (Placebo Comparator): 8 participants will be randomized in a 3:1 ratio to active or placebo. Study intervention will be administered orally once. Randomization to each SAD cohort will be done in a staggered manner; initially 2 sentinel participants (1 active and 1 placebo) will be randomized and dosed and after a safety evaluation period after the dose without clinically significant adverse events (AEs) and investigator approval, then, 6 additional participants will be randomized and dosed (5 active and 1 placebo) at the discretion of the Investigator according to the randomization schedule
  Interventions: Drug: Placebo
- Experimental Part 2: Active SPG302 to be administered to healthy volunteers (MAD) (Experimental): 8 participants will be randomized in a 3:1 ratio to active or placebo. Participants will receive study intervention QD over 5 days and will be discharged on Day 6. A follow-up safety visit will be conducted on Day 12 (±3 days).
  Interventions: Drug: SPG302
- Placebo Comparator Part 2: Placebo comparator to be administered to healthy volunteers (MAD) (Placebo Comparator): 8 participants will be randomized in a 3:1 ratio to active or placebo. Participants will receive study intervention QD over 5 days and will be discharged on Day 6. A follow-up safety visit will be conducted on Day 12 (±3 days).
  Interventions: Drug: Placebo
- Experimental Part 3: Active SPG302 to be administered to participants with ALS (Experimental): Participants with ALS will be randomized to receive SPG302 or placebo at a 3:1 ratio. Study intervention will be administered QD over 28 days. A follow-up safety visit will be conducted 30 days after last dose (±7 days). Participants who complete Part 3 may be offered to participate in an open-label extension.
  Interventions: Drug: SPG302
- Placebo Comparator Part 3: Placebo comparator to be administered to participants with ALS (Placebo Comparator): Participants with ALS will be randomized to receive SPG302 or placebo at a 3:1 ratio. Study intervention will be administered QD over 28 days. A follow-up safety visit will be conducted 30 days after last dose (±7 days). Participants who complete Part 3 may be offered to participate in an open-label extension.
  Interventions: Drug: Placebo
- Experimental Part 3: Open Label Extension - Active SPG302 administered to participants with ALS (Experimental): Participants with ALS will be randomized to receive SPG302 or placebo at a 3:1 ratio. Study intervention will be administered QD over 28 days for up to 3 cycles in the USA and up to 12 cycles in Australia. A follow-up safety visit will be conducted 30 days after last dose (±7 days).
  Interventions: Drug: SPG302

INTERVENTIONS:
Drug: SPG302 — synthetic small molecule
  Arms: Experimental Part 1: Active SPG302 to be administered to healthy volunteers (SAD); Experimental Part 2: Active SPG302 to be administered to healthy volunteers (MAD); Experimental Part 3: Active SPG302 to be administered to participants with ALS; Experimental Part 3: Open Label Extension - Active SPG302 administered to participants with ALS
Drug: Placebo — Placebo
  Arms: Placebo Comparator Part 1: Placebo comparator to be administered to healthy volunteers (SAD); Placebo Comparator Part 2: Placebo comparator to be administered to healthy volunteers (MAD); Placebo Comparator Part 3: Placebo comparator to be administered to participants with ALS

SUMMARY:
The first-in-human Phase 1 study described herein will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SPG302 in healthy volunteers and ALS participants

DETAILED DESCRIPTION:
This study is a Phase 1 randomized, double-blind, placebo-controlled, single, and multiple ascending dose study in HV with food effect cohort, and a repeat dose expansion cohort(s) in participants with ALS.

The study consists of 3 parts, as follows:

* Part 1: SAD in HV with up to 6 cohorts including a food effect cohort.
* Part 2: MAD over 5 days in HV with up to 5 cohorts
* Part 3: ALS cohorts with once daily (QD) dosing over 28 day cycles

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Must be in good health with no significant medical history
* Clinical laboratory values within normal range or < 1.2 times ULN
* BMI 18-32 (inclusive)
* Contraceptive use by men or women consistent with local regulations
* Able and willing to provide written informed consent

Exclusion Criteria:

* Any physical or psychological condition that prohibits study completion
* Known cardiac disease
* Active or history of malignancy in the past 5 years
* Serious infection within 1 month of screening
* Acute illness within 30 days of Day 1
* Surgery, bone fracture, or major musculoskeletal injury in the past 3 months
* History of suicidal behavior or suicidal ideation
* Active cigarette smokers and users of nicotine-containing products
* HIV, hepatitis B and hepatitis C positive
* SBP >140 or <90
* DBP >90 or <40
* HR <40 or >100
* QTcF >450ms, cardiac arrhythmia, or clinically significant abnormal ECG
* Prescriptions, over-the-counter, or herbal medication within 7 days
* Vaccines within 14 days
* Other investigational products within 30 days
* Blood donation within 30 days
* Plasma donation within 7 days
* Pregnant or breastfeeding
* Otherwise unfit, on metabolic-altering lifestyle/diet, positive urine drug screen or intake of alcohol or caffeine-containing products

ALS Cohort Inclusion Criteria:

* Age 18-80
* ALS TRICALS risk score
* Stable dose of standard of care treatment
* Contraception use by men or women consistent with local regulations
* Able and willing to provide written informed consent

ALS Cohort Exclusion Criteria:

* Underlying physical or psychological condition prohibiting study completion
* Known cardiac disease
* Active or history of malignancy in the past 5 years
* Serious infection within 1 month of screening
* Acute illness within 30 days of Day 1
* History of suicidal behavior or suicidal ideation
* Active cigarette smokers and users of nicotine-containing products
* Neurodegenerative disease
* External respiratory support or supplemental oxygen requirement
* HIV, hepatitis B and hepatitis C positive
* SBP >140 or <90
* DBP >90 or <40
* HR <40 or >100
* QTcF >450ms, cardiac arrhythmia, or clinically significant abnormal ECG
* Vaccines within 14 days
* Other investigational products within 30 days
* Blood donation within 30 days
* Plasma donation within 7 days
* Pregnant or breastfeeding
* Otherwise unfit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in healthy volunteers (SAD cohort) | 7 days
  • Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
Safety and tolerability in healthy volunteers (SAD food effect cohort) | 15 days
  • Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
Safety and tolerability in healthy volunteers (MAD cohort) | 12 days
  • Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
Safety and tolerability in participants with ALS | 60 days
  • Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Plasma pharmacokinetics of SPG302 in healthy volunteers (SAD cohort) | 7 days
  PK parameters of SPG302 on concentrations in plasma
Plasma pharmacokinetics of SPG302 in healthy volunteers (SAD food effect cohort) | 15 days
  Effects of food on SPG302 PK profile
Plasma pharmacokinetics of SPG302 in healthy volunteers (MAD cohort) | 12 days
  PK parameters of SPG302 on concentrations in plasma
Plasma pharmacokinetics of SPG302 in participants with ALS | 12mon
  PK parameters of SPG302 on concentrations in plasma
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12 mon
  Spirometry
Clinical efficacy measures of SPG302 in participants with ALS | 12 mon
  The Amyotrophic Lateral Sclerosis Functional Rating Scale-revised (ALSFRS-R).

OTHER OUTCOMES:
Effect of repeated dosing of SPG302 on electroencephalogram in healthy volunteers (MAD cohort) | 12 mon
  Change from baseline in EEG parameters
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12 mon
  Number of respiratory complications
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12 mon
  Spirometry
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12 mon
  TMS
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12 mon
  EEG
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12 mon
  Change in Nocturnal Pulse Oximetry
Clinical outcomes of multiple oral doses of SPG302 in participants with ALS | 12mon
  Edinburgh Cognitive and Behavioural ALS Screen (ECAS)
Effect of SPG302 on proteins and biomarkers in participants with ALS | 12mon
  Multiple protein and immunological biomarkers
The effect of SPG302 on protein(s) and biomarkers | 12mon
  Change from baseline in the analysis of Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Ofer M Gonen, MD, Principal Investigator — Nucleus Network (for healthy volunteers); David Schultz (ALS site), MD, Principal Investigator — Finders Medical Center (ALS); Robert Henderson (ALS site), MD, Principal Investigator — Royal Brisbane Hospital (ALS); Dominic Rowe, MD, Principal Investigator — Macquarie Hospital
Locations (4):
- Australia (4):
  - Macquarie University, North Ryde, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical center, Adelaide, South Australia
  - Nucleus Melbourne (healthy volunteers), Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No